### **Informed Consent Form**

Study Title: TeamTRACS Pilot (CTSI)

ClinicalTrials.gov ID (NCT number): NCT05370157

Document Date: January 18, 2023

#### CONSENT TO ACT AS A PARTICIPANT IN A RESEARCH STUDY

Improving Teamwork in Rural Child Advocacy Centers: A Hybrid Effectiveness-Implementation Trial of TeamTRACS

#### **Principal Investigator:**

Elizabeth A. McGuier, Ph.D. Assistant Professor of Psychiatry University of Pittsburgh 3811 O'Hara Street, Pittsburgh, PA 15213 (412) 246-5895 millerea3@upmc.edu

**Source of Support:** This study is funded by the Clinical and Translational Science Institute (CTSI) at the University of Pittsburgh.

#### What is this study about and why is it being done?

We are conducting a research study to evaluate the effects of TeamTRACS (<u>Team Training in Roles, Awareness, Communication, and Support</u>). TeamTRACS is a team training intervention designed to enhance and sustain healthy team functioning in Child Advocacy Centers (CACs). In this study, CACs will be randomized to TeamTRACS or a waitlist comparison. CACs randomized to the waitlist will receive TeamTRACS after completing the study. Our goals are to 1) test the effects of TeamTRACS on knowledge, skill use, and team functioning, and 2) assess the feasibility of a self-guided implementation approach.

#### Who is being asked to take part in this research study?

This study is recruiting CAC staff and multidisciplinary team members at participating CACs. We expect up to 200 individuals may participate.

#### What activities are part of the study?

- All team members will be invited to participate in TeamTRACS at their CAC.
- All team members will be invited to complete brief online surveys (<30 minutes) at the beginning of the study and 3 months later. Team members will also provide feedback immediately after participating in TeamTRACS. The surveys will assess different aspects of teamwork and perceptions of the training.
- Some team members will be invited to participate in individual qualitative interviews. We will conduct interviews about the multidisciplinary team at the beginning of the study and 3 months later. We will also conduct monthly interviews about the process of implementing TeamTRACS.
- CAC staff will be asked to report attendance at case review meetings and any changes in team members (e.g., turnover, addition of new members). CAC directors at the 4 CACs randomized to TeamTRACS will be asked to share documents created during the implementation process (e.g., worksheets, action plans, team goals).

#### How long will the study last?

Participants will be involved in the study for approximately 8 months and no more than 1 year.

#### Do I have to participate?

No. Your participation in this study is entirely voluntary. Whether or not you participate in this research study will not impact your employment, nor will your decision affect your current or future relationships with the University of Pittsburgh, UPMC or its affiliated health care providers, or health care insurance providers. The investigators are available to answer any questions you may have about the study.

What are the possible risks and benefits of participating in this research study? The risks to you are believed to be minimal and no greater than those experienced in daily life. It is possible that you may experience some inconvenience or discomfort when completing the surveys and/or interviews. You may skip any questions you prefer not to answer. You will be promptly notified if any new information we learn during this research study may cause you to change your mind about continuing to participate.

Participation does not provide any direct benefits to you. Your decision about participation will not impact your employment. Participation in this study may encourage you to reflect on team functioning, which may lead to improvements in team functioning, work performance, and outcomes for the children and families you serve. Team members who participate in TeamTRACS may increase their knowledge and use of teamwork skills. The information we obtain from you and others may help us learn how to better support CAC multidisciplinary teams.

#### Will I be paid if I take part in this research study?

Yes. You will receive \$20 for completing the pre-training survey, \$20 for completing the post-training survey, and \$30 for each completed qualitative interview. If you receive more than \$100 from this research study, you will be asked to provide your social security number, and your name, address, and social security number will be released to the Accounting Office. You do not have to provide your social security number if you do not wish to. If the total reimbursement for your participation in research is greater than \$600 in a year, this will be reported to the Internal Revenue Service (IRS) as income.

#### Are my responses private?

- The research team will do everything possible to ensure your responses are
  private. You can complete online surveys in a time and place of your choosing to
  maximize privacy. For interviews, the interviewer will be in a private office and
  verify that you are in a private location where you are unlikely to be interrupted
  prior to starting the interview.
- Only the research team will have access to your data. Survey responses and
  interview recordings will be labeled with ID numbers that do not identify you and
  stored on secure, password-protected servers. The information linking these
  case numbers with your identity will be kept separate from the research records.

- Individual responses will not be shared, and your identity will not be revealed in any description or publications of this research. Other researchers may ask to review and use data from this study for their own research. To protect your privacy, we will carefully consider each request and will remove anything that could identify you before sharing any data with other researchers.
- No individual information will be shared with your employer or leadership.
   Although every reasonable effort has been taken, confidentiality during Internet communication activities cannot be guaranteed and it is possible that additional information beyond that collected for research purposes may be captured and used by others not associated with this study.

## Who will have access to my identifiable information related to my participation in this study?

In addition to the investigators listed on the first page of this consent form and their research staff, the following individuals will or may have access to identifiable information related to your participation in this research study:

- Authorized representatives of the University of Pittsburgh Office of Research Protections may review your identifiable research information for the purpose of monitoring the appropriate conduct of this research study.
- In unusual cases, the investigators may be required to release your identifiable research information in response to an order from a court of law. If the investigators learn that you or someone with whom you are involved is in serious danger or potential harm, they will need to inform the appropriate agencies, as required by Pennsylvania law.
- The fact that you are participating in a research study may also be known to individuals involved in administrative activities associated with the conduct of the study.

# For how long will the investigators be permitted to use and disclose identifiable information related to my participation in this research study?

Per University of Pittsburgh policy, research records will be maintained for at least 7 years after the final reporting or publication of a project.

May I withdraw, at a future date, my consent to participate in this research study? You may withdraw your consent for your participation in this study at any time. Any information recorded for or resulting from your participation in this study prior to the date that you formally withdrew your consent may continue to be used as described above. To formally withdraw your consent for your participation in this research study you should provide a written and dated notice of this decision to the study's principal investigator at the address listed at the top of this form. Your decision to withdraw your consent for participation in this research study will not impact your employment, nor will your decision affect your current or future relationships with the University of Pittsburgh, UPMC or its affiliated health care providers, or health care insurance providers.

If I agree to take part in this research study, can I be removed from the study without my consent?

It is possible that you may be removed from the research study by the investigators if you are no longer part of the participating multidisciplinary team, you are no longer able to participate, and/or if you do not follow the instructions given by the investigator and the research team. Any identifiable research information recorded for, or resulting from, your participation in this research study prior to the date that you were removed from the study may continue to be used and disclosed by the investigators for the purposes described above.

May I be contacted about possible participation in future research studies? You may be contacted in the future about possible research studies for which you might be eligible. You are under no obligation to participate in any future study.

#### Who do I contact if I have questions about the study?

You can contact the principal investigator listed at the top of this form via phone or email with any questions. If you have any questions about your rights as a research subject or wish to talk to someone other the research team, please call the University of Pittsburgh Human Subjects Protection Advocate toll-free at 866-212-2668.

#### **VOLUNTARY CONSENT**

If you agree to participate, please choose the "I consent to participate" option below. Choosing this option implies that you have read the information on this form, your current questions have been answered, that you understand that you are encouraged to ask questions about any aspect of this research study, and that such future questions will be answered by a qualified individual or by the investigator(s) listed at the top of this consent document at the telephone number(s) given. Your consent further indicates that you understand that you may contact the Human Subjects Protection Advocate of the IRB Office, University of Pittsburgh (1-866-212-2668) to discuss problems, concerns, and questions; obtain information; offer input; or discuss situations in the event that the research team is unavailable. You may print a copy of this page as a record of your consent to participate.

| If you choose not to participate in this study, please select the "I do not consent to |
|---|
| participate" option and close your web browser. |
| □ I consent to participate |
| □ I do not consent to participate |
| · · |